CLINICAL TRIAL: NCT02527577
Title: Analgesia by Transversus Abdominis Plane Nerve Block in Patients Undergoing Liver Resection
Acronym: BLOC-TAP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulties to recruit patients
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0908127; 2009-017768-18 (EudraCT Number); A100140-28 (Other: AFSSAPS)
Record Dates: First submitted 2015-08-14; First posted 2015-08-19 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-07

CONDITIONS: Liver Cancer, Adult
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ropivacaïne chlorhydrate monohydrate (Experimental)
  Interventions: Drug: RopivacaIne chlorhydrate
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RopivacaIne chlorhydrate — 3mg/kg injection Hour (H) 0, H12 ; H24, H36 ; H48
  Other Names: 3mg/kg
  Arms: ropivacaïne chlorhydrate monohydrate
Drug: Placebo — injection Hour (H) 0, H12 ; H24, H36 ; H48
  Other Names: NaCl 0,9%
  Arms: placebo

SUMMARY:
The indications liver cancer surgery currently booming due to the increase in surgical techniques and instruments for a more secure resection of liver tissue with a significant reduction in bleeding or surgical complications. This allowed to expand surgical indications in the most fragile patients so assuming optimized anesthetic care.

So far, the technique of analgesia reference to this surgery remains administration of morphine analgesia via a device controlled by the patient (PCA) for epidural analgesia is against-indicated because of induced bleeding disorders by surgery.

Rafi then McDonnell in 2007 have described a new technique of loco regional anesthesia, the abdomen of the Transversus Abdominis Plane (TAP) nerve block(TAP), which allows selective anesthesia of the abdominal wall. But parietal pain related muscular and nervous sagging surgical approach represent a significant share of post operative pain.

This study proposes an evaluation of the abdomen transverse blocks in hepatectomy.

ELIGIBILITY:
Inclusion Criteria:

* hepatectomy or segmentectomy

Exclusion Criteria:

* Sepsis uncontrolled current
* Overdose in anticoagulant during general anesthesia
* Thrombocytopenia <50 g / dl
* Severe renal impairment: Cockcroft <30 ml / min
* history of ventricular arrhythmia serious unexplained .*
* Allergy to local anesthetics of the amide
* Contraindication to remifentanil and morphine
* Hypovolemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2010-04; Primary Completion 2014-09 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
consumption of morphine over the first 48 hours postoperative. | at 48 hours postoperative

SECONDARY OUTCOMES:
pharmacokinetic of ropivacaine (plasma concentrations) | 1, 2, 3, 6, 10, 24, 36, 48 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: carine.labruyere@chu-st-etienne.fr MOLLIEX, MD PhD, Principal Investigator — CHU de SAINT-ETIENNE
Locations (1):
- CHU de SAINT-ETIENNE, Saint-Etienne, France